CLINICAL TRIAL: NCT00000445
Title: Effectiveness of Naltrexone in a Community Setting
Brief Title: Use of Naltrexone in a Clinical Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NIAAABRA11747
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-07

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

INTERVENTIONS:
Drug: naltrexone (Revia)

SUMMARY:
This 12-week trial will compare individuals receiving naltrexone or placebo plus substance abuse counseling therapy versus those receiving only substance abuse counseling therapy in a rural, nonacademic setting. A followup period of 12 months is included. The effect on service utilization and the cost of the addition of naltrexone to treatment services for alcohol dependence also will be assessed. The study will expand existing research concerning the effectiveness of naltrexone in clinical trials versus a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol dependence (within the past 3 months).
* Meets criteria for another substance use disorder (except narcotic dependence) but must identify alcohol as the primary substance of abuse.
* Must be able to provide an informed consent.
* Consent to random assignment and be willing to commit to possible medication treatment and research follow-up.
* Must be eligible for treatment at the Dorchester Alcohol and Drug Commission.

Exclusion Criteria:

* Meets criteria for opiate dependence.
* Clinically significant medical problems such as collagen-vascular disease, cardiovascular, renal, gastrointestinal or endocrine problem that would impair participation or limit medication ingestion.
* Hepatocellular disease.
* Women who are pregnant, nursing, or not practicing an effective means of birth control.
* Currently being prescribed naltrexone.
* Known sensitivity or allergy to naltrexone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Drug and Alcohol Programs, Medical University of South Carolina, Charleston, South Carolina, United States